CLINICAL TRIAL: NCT02662400
Title: Assessment of Insulin Sensitivity and β Cell Function by Clamps Studies After Stem Cell Transplantation in T2DM
Brief Title: Assessment of Insulin Sensitivity and β Cell Function by Clamps Studies
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, Profeesor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNCs IN Diabetes
Record Dates: First submitted 2016-01-10; First posted 2016-01-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MNCs GROUP (Experimental): Patients with Type 2 Diabetes mellitus
  Interventions: Biological: MNCs

INTERVENTIONS:
Biological: MNCs — 200 - 300 ml of bone marrow will be aspirated and layered on density gradient medium (Ficoll - hypaque ) and stem cells will be separated. Separated mono nucleated cells will injected into superior pancreatico duodenal artery. Patients will be urged to monitor and document blood glucose readings for next 6 months. Glucagon stimulated C - peptide HYPERGLYCEMIC CLAMP FOR ASSESSMENT OF BETA CELL FUNCTION , AND EUGLYCEMIC CLAMP TO ASSESS INSULIN SENSITIVITY .Homeostasis Model of Assessment - Insulin Resistance and Beta cell function ,HbA1c, lipid profile and biochemistry will be done at baseline and 6 months

SUMMARY:
India is the "Diabetes Capital of the World" with 41 million Indians having diabetes i.e. every fifth diabetic in the world is an Indian. Type 2 Diabetes Mellitus (T2DM) constitutes the major chunk of diabetes and has insulin resistance as the hallmark feature in the pathogenesis. However, with the progression of the disease the insulin resistance becomes stable whereas β - cell function shows a gradual decline due to its ongoing apoptosis. This ultimately leads to inability of the β - cells to cope up with the increased demand of insulin caused due to insulin resistance and manifests as hyperglycemia. As β - cell failure is progressive and inexorable, as demonstrated in United Kingdom Prospective Diabetes Study, most of the patients with T2DM would eventually require insulin and it would be difficult to achieve to attain a strict glycemic control . It is well known that diabetes related complications which account for morbidity and mortality in this disease can be prevented or delayed by strict glycemic control. However, even with intensive insulin therapy it has been shown that glycemic control can never be perfect with patients exhibiting hyperglycemia or hypoglycemia during 24 hour glucose profile. Also insulin therapy is not physiological as there is no hepatic "first - pass" metabolism of insulin which is required for halting the hepatic glucose output, which is responsible for fasting hyperglycemia. This led the researchers to evolve various strategies of β - cell replacement therapy e.g. pancreatic transplantation and islet cell transplantation. Initially the results of islet cell transplantation were dismal but after the induction of glucocorticoid free immunosuppressive therapy and the use of adequate number of islet cells from multiple donors, the results of islet cell transplantation have been better. However, islet cell transplantation has its own limitations viz insufficient supply, being technically demanding and requirement of lifelong immunosuppressive therapy in the recipient.

DETAILED DESCRIPTION:
The shortcomings can be overcome by the use of stem cells which is an inexhaustible source of β -cells. Stem cells are primitive cells capable of differentiating into mature cells of the body of various lineages. Stem cells can be obtained from various sources like blastocyst (embryonal stem cells), umbilical cord or bone marrow. There is an evidence to suggest that stem cell transplantation can lead to improvement in pancreatic endocrine function and improvement in glycemic control in diabetic mice through various mechanisms such as transdifferentiation or regeneration of endothelial cell in the damaged islets which in turn lead to regeneration of islet cells by paracrine action. However, till date there is no study that demonstrates that stem cell therapy can be effective in patients with T2DM for their glycemic control.

The investigators propose to carry out autologous bone marrow - derived stem cell transplantation (ABMSCT) in patients of T2DM, obtained from their own bone marrow and its superselective injection into the gastroduodenal artery after purification without any immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* Failure to triple oral hypoglycemic agent and on stable doses of insulin for at least 3 months.
* On vildagliptin,pioglitazone and metformin for at least 3 months along with Insulin to maintain euglycemia.
* HbA1c < 7.5%.
* Insulin requirement ≥0.4 IU/kg/d.
* GAD antibody negative status.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or secondary diabetes.
* Patients with serum creatinine > 1.5 mg/dl.
* Abnormal liver function tests (defined as value of transaminases > 3 times the upper value of normal or serum bilirubin higher than normal for the reference value for the laboratory).
* History of cholecystitis/ cholelithiasis/cholecystectomy.
* Seropositivity for HIV, HBsAg and hepatitis C virus (HCV).
* History of myocardial infarction or unstable angina in the previous 3 months.
* History of malignancy.
* Patients with active infections.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in insulin sensitivity after stem cell transplantation | 6 months
  Stem cells will be transplanted in patients with T2DM. Pre and Pro stem cell transplantation Insulin sensitivity(pmol/l) will be assessed by euglycemic clamp .

SECONDARY OUTCOMES:
Improvement in β cell function after stem cell transplantation | 6 months
  Stem cells will be transplanted in patients with T2DM. Pre and Pro stem cell transplantation β cell function(nmol/L) will be assessed by hyperglycemia clamp .

CONTACTS AND LOCATIONS:
Overall Officials: anil Bhansali, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhansali A, Asokumar P, Walia R, Bhansali S, Gupta V, Jain A, Sachdeva N, Sharma RR, Marwaha N, Khandelwal N. Efficacy and safety of autologous bone marrow-derived stem cell transplantation in patients with type 2 diabetes mellitus: a randomized placebo-controlled study. Cell Transplant. 2014;23(9):1075-85. doi: 10.3727/096368913X665576. PMID 23561959